CLINICAL TRIAL: NCT06266845
Title: Efficacy of Gamification With Escape-Room for Arrhythmia Identification in Critical Patients: an Experiment With Nursing Undergraduates
Brief Title: Efficacy of Gamification With Escape-Room for Arrhythmia Identification in Critical Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Brasilia (Other)
Responsible Party: Principal Investigator, Marcia Cristina da Silva Magro, Clinical Professor, University of Brasilia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 76082423.1.0000.8093
Record Dates: First submitted 2024-01-27; First posted 2024-02-20 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Arrythmia; Health Education; Escape-Room
MeSH Terms: conditions — Arrhythmias, Cardiac; Health Education

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Knowledge Test (Other)
  Interventions: Behavioral: In-person Escape Room; Behavioral: Virtual Escape-Room
- Knowledge Test Satisfaction and Self-Confidence Scale (Other)
  Interventions: Behavioral: In-person Escape Room; Behavioral: Virtual Escape-Room
- Perceived Gains Scale and DASS-21 (Depression, Anxiety, and Stress Scale-21) (Other)
  Interventions: Behavioral: In-person Escape Room; Behavioral: Virtual Escape-Room

INTERVENTIONS:
Behavioral: In-person Escape Room — The in-person escape room will be conducted in the nursing laboratory of a Higher Education Institution (HEI), equipped with a high-fidelity mannequin to simulate a critical patient and create a realistic environment. Participants will be divided into groups, with one group entering at a time as requested. During the in-person escape room, participants will interact with the patient mannequin, hospital equipment and devices, as well as with objects and clues in the environment. The game duration will be 30 minutes to ensure equal conditions among participants and prevent time distortions. Interactions and participants' performance will be recorded by the facilitator, guiding the feedback.
Behavioral: Virtual Escape-Room — The virtual escape room will be conducted in a classroom of an HEI, utilizing an online platform that allows the virtual reproduction of the game. Each group will have access to a tablet or computer to participate in the game provided by the researcher. During the game, participants will interact with the platform interface and solve challenges to escape the virtual room within 30 minutes. Thus, each group will have a maximum of 30 minutes to complete the escape room, ensuring equal conditions among participants. Records of interactions and participant performance will be logged for later analysis and feedback.

SUMMARY:
Introduction: Health education provided through the escape-room is still a recent approach in educational methodology and tends to be a strategy that benefits nursing students, particularly in gaining knowledge and skills. However, few studies have explored the use of both in-person and virtual escape-room as an educational methodology in nursing. Objective: To assess the effectiveness of the gamification strategy through the in-person escape-room model compared to the virtual model in enhancing cognitive and affective competencies for recognizing cardiac arrhythmias in critical care patients within the nursing field. Method: A randomized clinical trial to be conducted with nursing students from higher education institutions in the Federal District, Brazil. Students will undergo a theoretical class on cardiac arrhythmias in critical patients and will then be randomized to experience either the in-person or virtual escape-room scenario. Knowledge tests, the Depression, Anxiety, and Stress Scale, Satisfaction and Self-confidence Scale in nursing management learning, and perceived gains will be administered pre and post-intervention. Results with p≤0.05 will be considered significant. Expected Results: It is anticipated that this study will contribute to the enhancement and broadening of cognitive and affective competencies in nursing students, improving the quality of care through an active educational strategy like the escape-room, and consequently reducing costs for the Unified Health System by minimizing errors in recognizing clinical changes in critical patients. Additionally, the study aims to address gaps in understanding the use of educational escape-rooms in the field of nursing.

ELIGIBILITY:
Inclusion Criteria:

* Students enrolled in the undergraduate nursing program who have successfully completed the course related to adult and elderly health.

Exclusion Criteria:

* Healthcare professionals, including those participants who, at any point during the research stages, choose to withdraw or who have not completed/participated in one of the study phases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the feelings of stress and anxiety among nursing students after experiencing the in-person and virtual escape-room combined with an interactive lecture | 3 months
  The Depression, Anxiety, and Stress Scale (DASS-21) will be necessary to assess the impact of the intervention on the stress experienced by students during the process. The scale consists of 21 items, with seven items in each of the three scales (depression, anxiety, and stress). The minimum and maximum scores for each subscale are determined by the sum of the values assigned to the corresponding items. Generally, for each of the three subscales, the minimum possible score is 0, indicating the absence of symptoms, while the maximum score varies depending on the intensity of the responses provided by participants to specific items. For example, on a scale of 0 to 21 for each subscale, a higher score suggests higher levels of depression, anxiety, or stress.
Perceived Gains Scale | 3 months
  Another instrument that will be used in the study is the Perceived Gains Scale, which consists of 25 items with 5 response options: Improved immensely; improved considerably; improved slightly; stayed the same; got worse. In this scale, the different variables identify students' perceptions of the gains achieved through their experience with high-fidelity patient mannequins at the cognitive level.
Student Satisfaction and Self-Confidence in Learning | 3 months
  The "Student Satisfaction and Self-Confidence in Learning" Scale was developed to measure individuals' satisfaction and self-confidence acquired through high-fidelity simulations. This instrument has been validated in Brazil and will be used in the present study following the intervention. The scale consists of 26 items, organized into five factors: the usefulness and effectiveness of teaching methods, the provision of didactic materials and activities, the quality of teaching provided by the facilitator, self-confidence in learning, and student responsibility for their own learning. Participants indicate their level of agreement with each item on a five-point scale, ranging from "strongly disagree" to "strongly agree." The closer to 5, the higher the level of satisfaction with learning and self-confidence.

CONTACTS AND LOCATIONS:
Locations (1):
- Alberto Augusto Martins Paiva, Brasília, Federal District, Brazil

IPD SHARING:
Plan to Share IPD: No